CLINICAL TRIAL: NCT02326662
Title: Safety and Efficacy of Autologous Neural Stem Cell Transplantation in Patients With Traumatic Spinal Cord Injury
Brief Title: Neural Stem Cell Transplantation in Traumatic Spinal Cord Injury
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government)
Collaborators: Novagenesis Foundation (Unknown); Ophiuchus Technologies AG (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: FMBA OPH1
Record Dates: First submitted 2014-11-30; First posted 2014-12-29 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; neural stem cells; paraplegia; transplantation
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Paraplegics Acute (Experimental): Acute [1-6 mo.] patients (paraplegics) with major complete traumatic spinal cord injury that will undergo autologous neural stem cell transplantation including RMx Biomatrix as scaffold for the stem cells as needed Intervention: Autologous Stem Cell Transplantation with a 3D biomatrix.
  Interventions: Biological: Autologous Stem Cell Transplantation
- Paraplegics Sub-chronic (Experimental): Sub-chronic [6-12 mo.] patients (paraplegics) with major complete traumatic spinal cord injury that will undergo autologous neural stem cell transplantation including RMx Biomatrix as scaffold for the stem cells as needed Intervention: Autologous Stem Cell Transplantation with a 3D biomatrix.
  Interventions: Biological: Autologous Stem Cell Transplantation
- Paraplegics Chronic (Experimental): Chronic [1- 5 years]) patients (paraplegics) with major complete traumatic spinal cord injury that will undergo autologous neural stem cell transplantation including RMx Biomatrix as scaffold for the stem cells as needed.
  Intervention: Autologous Stem Cell Transplantation with a 3D biomatrix.
  Interventions: Biological: Autologous Stem Cell Transplantation
- Tetraplegics Acute (Experimental): Acute [1-6 mo.] patients (tetraplegics) with major complete traumatic spinal cord injury that will undergo autologous neural stem cell transplantation including RMx Biomatrix as scaffold for the stem cells as needed Intervention: Autologous Stem Cell Transplantation with a 3D biomatrix.
  Interventions: Biological: Autologous Stem Cell Transplantation
- Tetraplegics Sub-chronic (Experimental): sub-chronic [6-12 mo.] patients (tetraplegics) with complete traumatic spinal cord injury that will undergo autologous neural stem cell transplantation including RMx Biomatrix as scaffold for the stem cells as needed.
  Intervention: Autologous Stem Cell Transplantation with a 3D biomatrix.
  Interventions: Biological: Autologous Stem Cell Transplantation
- Tetraplegics Chronic (Experimental): Chronic [1- 5 years]) patients (tetraplegics) with major complete traumatic spinal cord injury that will undergo autologous neural stem cell transplantation including RMx Biomatrix as scaffold for the stem cells Intervention: Autologous Stem Cell Transplantation & Biomatrix
  Interventions: Biological: Autologous Stem Cell Transplantation

INTERVENTIONS:
Biological: Autologous Stem Cell Transplantation — Autologous neural stem cell transplantation Stem Cell Transplantation by intraspinal and intrathecal injection with 3D matrix as needed

SUMMARY:
This research investigates the use of autologous neural stem cells in patients with complete traumatic spinal cord injury.

DETAILED DESCRIPTION:
The aim of this study is to evaluate Mesenchymal Stem Cells [MSC]-derived autologous neural stem cells transplantation as a safe and potentially beneficial treatment for patients with traumatic spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years old
* Traumatic spinal cord injury at the neck, thoracic or lumbar level
* Classification ASIA A and B with no significant further improvement with physical therapy/rehabilitation
* A score of less than 200 in the 324-point ASIA scale
* Injury duration 1 month to 5 years

Exclusion Criteria:

* An advanced, severe, or unstable disease of any type that may interfere with primary and secondary variable evaluations, including any medical condition that could be expected to progress, recur, or change to such an extent that it may bias the assessment of the clinical or mental status of the patient to a significant degree or put the patient at special risk (e.g., severe liver or kidney disease, malignancies/cancer)
* Immune system disorder or dysfunction
* Any major/serious infections up to 2 months prior to inclusion
* A disability that may prevent the patient from completing all study requirements (e.g., blindness, deafness, severe language difficulty)
* A current diagnosis of active, uncontrolled peptic ulceration within the last three months
* A current diagnosis of acute, severe, or unstable asthmatic conditions [e.g., severe chronic obstructive pulmonary disease (COPD)]
* Participated in any other investigational trial within 4 weeks of initial screening and within 7 weeks of study entry
* History of regular alcohol intake or drug abuse in the previous 3 months and not able to sustain from alcohol intake during the trial Cardiovascular
* A current diagnosis of severe or unstable cardiovascular disease
* A current diagnosis of sick-sinus syndrome or conduction deficits (e.g., sino-atrial block, second or third degree atrio-ventricular block)
* A current diagnosis of uncontrolled atrial fibrillation (>100 bpm)
* A current diagnosis of moderate to severe heart failure [New York Heart Association (NYHA), Class III or more]
* A myocardial infarction (MI) known to have occurred within the last 3 months
* A current diagnosis of severe or unstable angina
* Vital signs (supine) outside the following ranges
* Systolic blood pressure below 90 or above 160 mmHg
* Diastolic blood pressure below 55 or above 95 mmHg
* Radial pulse below 50 or above 100 bpm CNS related
* A recent history of up to one year or currently diagnosed with cerebrovascular disease (e.g., stroke transient ischemic attacks, aneurysms)
* A current diagnosis of any primary neuro-degenerative disorder [e.g., Huntington's disease, Parkinson's disease etc.]
* A current diagnosis of an active, uncontrolled seizure disorder Psychiatric
* A current DSM-IV diagnosis of major depression
* Any other DSM-IV Axis 1 diagnosis that may interfere with the response of the patient to study medication, including other primary degenerative dementia, schizophrenia, or bipolar disorder Laboratory abnormalities
* Clinically significant abnormalities in routine laboratory examinations (hematology, electrolytes, biochemistry, liver and kidney function tests, urinanalysis) Concomitant therapy
* Previous stem cell treatment
* Ingested any of the following substances
* An investigational drug during the past 6 months
* A drug or treatment known to cause effect on the central nervous system [CNS] during the past four weeks
* A drug or treatment known to cause major organ system toxicity during the past four weeks
* Anticholinergic drugs at baseline
* Medication for Parkinson's disease at baseline (e.g., selegiline, levodopa, amantadine, dopamine agonists, COMT inhibitors)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-07; Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility and safety of autologous Neural Stem Cell transplantation in patients with complete traumatic spinal cord injury as measured by reported side effects and surgery procedure | 24 months
  Side effects is recorded by the hospital staff, in the CRF and by the patient. Surgery procedure is documented by video and standard recording

SECONDARY OUTCOMES:
324-point ASIA and other scoring incl. muscle control and voluntary movement and improvement of sphincters control | 3, 6,12, 24 months and 3 year follow-up
  Change from Baseline in ASIA Score. All patients are stable ASIA A.
MRI Scan of Spinal Cord | 3, 6,12, 24 months and 3 year follow-up
  Change from Baseline of Injury Area. All patients has spinal cord injuries visible on MRI

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Averyanov, MD, Principal Investigator — Federal Research Clinical Center FMBA of Russia
Locations (1):
- Federal Research Clinical Center FMBA of Russia, Moscow, Russia